CLINICAL TRIAL: NCT03521050
Title: LUKS-Leads Registry on Long-term Performance of ICD Leads
Status: Recruiting | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Richard Kobza, PD Dr. med., Luzerner Kantonsspital
Other Study IDs: 2016-02002
Record Dates: First submitted 2017-11-27; First posted 2018-05-11 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Defibrillators; Electrical Shock
MeSH Terms: interventions — Device Lead Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- implanted defibrillator lead: patients having an ICD implanted and having follow-up at the investigators center
  Interventions: Device: defibrillator lead

INTERVENTIONS:
Device: defibrillator lead — observation of long-term performance of defibrillator leads

SUMMARY:
All patients having an implantable cardiac defibrillator (ICD) implanted and having follow-up at the Cantonal Hospital Lucerne (LUKS), the investigator center, are included in this retrospective ICD lead registry from 2006 onwards. Data is collected prospectively from december 2016 onwards. After certain ICD-leads tended to fail early the investigators aimed for a registry monitoring our patient population with defibrillator leads and evaluating their long-term performance.

DETAILED DESCRIPTION:
All patients having an ICD implanted and having follow-up at the investigators center are included in this retrospective ICD lead registry from 2006 onwards. Data is collected prospectively from december 2016 onwards. After certain ICD-leads tended to fail early the investigators aimed for a registry monitoring our patient population with defibrillator leads and evaluating their long-term performance.

The following parameters will be measured during regular clinical controls: electronic impedances, threshold values, sensing values, battery performance, inadequate/adequate shock release und software problems

ELIGIBILITY:
Inclusion Criteria:

* all patients being implanted with a Defibrillator lead from 2006 onwards

Exclusion Criteria:

* documented refusal of data collection for scientific purposes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a clinical indication for an ICD
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
performance of lead impedance | regular clinical controls within 10 years
  electronic impedances in Ω
performance of lead threshold | during regular clinical controls within 10 years
  threshold values in V
performance of lead sensing | during regular clinical controls within 10 years
  sensing values in millivolt (mV)
lead parameters | during regular clinical controls within 10 years
  battery performance in %
performance of defibrillator | during regular clinical controls within 10 years
  inadequate/adequate shock release in numbers
control system of defibrillator | during regular clinical controls within 10 years
  software problems in numbers and descriptive

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kobza, MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Heart Centre, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No